CLINICAL TRIAL: NCT04097964
Title: Examining the Effectiveness of the FaCES Adolescent SBIRT Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Friends Research Institute, Inc. (Other)
Collaborators: Conrad N. Hilton Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 16743
Record Dates: First submitted 2019-09-19; First posted 2019-09-20 (Actual); Last update posted 2021-10-22 (Actual); Status verified 2021-10

CONDITIONS: Adolescent Health Services; Adolescent Behavior
Keywords: SBIRT
MeSH Terms: conditions — Adolescent Behavior | interventions — Crisis Intervention; Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FaCES Intervention (Experimental): Primary care providers will deliver anticipatory guidance for adolescents reporting no drug, alcohol or marijuana use in past year, an abbreviated brief intervention for adolescents who report using these substances one or twice in the past year, and a full brief intervention for adolescents who report using these substances monthly or weekly in the past year.
  Interventions: Behavioral: brief intervention
- Treatment as usual (Active Comparator): Usual care will be delivered by primary care providers during the clinic visit
  Interventions: Behavioral: treatment as usual

INTERVENTIONS:
Behavioral: brief intervention — 1 minute or less of anticipatory guidance will be provided for adolescents reporting no use in the past year, a 3-5 minute abbreviated brief intervention including raising the subject, asking more questions, and correcting misinformation will be provided for adolescents reporting substance use once or twice in the past year, and a 5-10 minute full brief intervention will be provided, including the above steps as well as assessing readiness and negotiating change and scheduling a follow-up to potentially include a referral to treatment will be provided to adolescents reporting monthly to weekly use in the past year.
  Arms: FaCES Intervention
Behavioral: treatment as usual — standard care conducted by primary care providers during clinic visits
  Arms: Treatment as usual

SUMMARY:
The study will utilize a stepped wedge cluster randomized design to examine the effectiveness of the full FaCES (Facilitating Change for Excellence in SBIRT) adolescent SBIRT change package. Primary care providers will be randomized as to when they receive training and begin delivery of FaCES with their 12 to 17 year old patients, which includes targeted feedback based on the patient's endorsed substance use level on the S2BI screening instrument.

DETAILED DESCRIPTION:
The study will utilize a stepped wedge cluster randomized design to examine the effectiveness of the full FaCES (Facilitating Change for Excellence in SBIRT) adolescent change package for 12 to 17 year old primary care patients. Primary care providers at two rural federally qualified health centers in New Mexico and Tennessee will be randomized as to when they receive training and begin delivering FaCES to their adolescent patients. FaCES includes targeted feedback based on the patient's endorsed substance use level on the S2BI screening instrument. Study participants will complete a baseline and follow-up assessment 3-months post study recruitment.

ELIGIBILITY:
Inclusion Criteria:

* Ages 12 to 17 years, inclusive
* Registered patient at one of the participating FQHCs
* Able and willing to provide informed consent

Exclusion Criteria:

* Inability to comprehend the assent form
* Parent/guardian declines consent

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1226 (Actual)
Dates: Start 2018-03-15 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
S2BI | 3 months
  S2BI score change

SECONDARY OUTCOMES:
ASSIST | 3 months
  The Alcohol, Smoking and Substance Involvement Screening Test
BSTAD | 3 months
  Brief Screener for Tobacco, Alcohol, and other Drug Use

CONTACTS AND LOCATIONS:
Overall Officials: Shannon G Mitchell, PhD, Principal Investigator — Friends Research Institute, Inc.
Locations (4):
- United States (4):
  - Hidalgo Medical Services, Lordsburg, New Mexico
  - Hidalgo Medical Services, Silver City, New Mexico
  - Lifespan Health, Adamsville, Tennessee
  - Lifespan Health, Savannah, Tennessee

IPD SHARING:
Plan to Share IPD: No